CLINICAL TRIAL: NCT05822960
Title: To Investigate the Effect of Far-infrared Radiation on Lower Extremity Acupoints on the Blood Circulation of Lower Extremities in Patients With Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202212028DINA
Record Dates: First submitted 2023-03-06; First posted 2023-04-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Arterial Disease
Keywords: hemodialysis; peripheral arterial occlusion disease; far-infrared radiation; lower extremity acupoints; ankle-brachial index; Edinburgh claudication questionnair
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: The dialysis day was W 1.3.5 as the control group and W 2.4.6 as the experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- far-infrared radiation on foot acupoints (Experimental): experimental group far-infrared radiation on foot acupoints during dialysis,during dialysis,, and the irradiation distance was 20 cm for 40 minutes each time for six months.
  Interventions: Device: far-infrared radiation
- The control group received general clinical routine care (No Intervention): no far-infrared radiation on foot acupoints

INTERVENTIONS:
Device: far-infrared radiation — far-infrared radiation on foot acupoints (Yinlingquan and Sanyinjiao acupoints) during dialysis
  Arms: far-infrared radiation on foot acupoints

SUMMARY:
This study intends to irradiate the acupoints of both lower extremities of hemodialysis patients with far-infrared therapeutic apparatus to explore its effect on foot blood circulation, peripheral artery occlusion disease (PAOD) symptoms and ankle-brachial index (Ankle-Brachial Index, ABI) value.

DETAILED DESCRIPTION:
After irradiating the lower extremity acupoints of hemodialysis patients with far-infrared rays, it is expected to improve the blood circulation of the lower extremities of hemodialysis patients, thereby improving the symptoms of indirect claudication and raising the ankle-brachial index to the normal range, and reducing the incidence of peripheral arterial disease in hemodialysis patients. The results of this study can provide an empirical reference for future clinical care.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients diagnosed with chronic renal failure in a hemodialysis unit and receiving hemodialysis for at least three months 2. Willing to participate in interventional treatment with far-infrared radiation 3. Willingness to cooperate with intervention measures and inspection time 4. Receive hemodialysis treatment three times a week

Exclusion Criteria:

1. There are contraindications for ABI examination (such as breast cancer lymph node dissection in the past), bilateral upper limb arteriovenous access, etc.), and a double- lumen dialysis venous catheter is placed in the groin
2. Bedridden or unable to walk
3. History of distal amputation, DVT, CABG s/p due to trauma, ischemia or infection
4. Consciously unclear and unable to cooperate
5. Patients with wounds from calf to instep

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Comparison of the "Edinburgh Claudication Questionnaire" and "ABI" after receiving far-infrared lower extremity acupoint irradiation therapy (investigators ) and general clinical care (participants) change assessed | intervention 1,2,3 and 6 month change is being assessed
  investigators :receiving far-infrared intervention;participants :general clinical care

SECONDARY OUTCOMES:
Comparison of basic data and disease characteristics distribution between the two groups | two groups before receiving far-infrared intervention (month 0)"change" is being assessed
  Demographic characteristics include: gender(boy or gril), age, education level, smoking history, presence/absence of exercise, and drinking; disease characteristics include(yes or no): years of dialysis(year), presence/absence of anticoagulant drugs(yes or no); disease history(yes or no): diabetes, hypertension, coronary artery disease disease, cerebrovascular disease The monthly routine inspection items in the hemodialysis room are designed,
To compare the "Edinburgh claudication questionnaire" and "ABI" before (month 0) receiving far-infrared lower extremity acupoint irradiation therapy and general clinical care | two groups before receiving far-infrared intervention (month 0)"change" is being assessed,
  In this study, used the Chinese version of the "Edinburgh Claudication Questionnaire" as a screening test for "intermittent claudication symptoms"; This study intends to use ABI-type equipment for measurement. Because hemodialysis patients have the limitation that the arm on the side of the arteriovenous fistula can not measure blood pressure, the modification is as follows Calculation method: ABI of left foot = systolic pressure of left posterior tibia ÷ systolic pressure of brachial artery without arteriovenous fistula;ABI of right foot is also calculated in the same way

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Yunlin Branch hemodialysis room, Huwei, Taiwan

IPD SHARING:
Plan to Share IPD: No